CLINICAL TRIAL: NCT06959251
Title: A Randomized, Placebo-controlled Clinical Trial Evaluating the Efficacy and Safety of Glycine and Magnesium+Thiamine Supplements, Alone or Combined, Administered for 6 Months to Patients With Primary Ciliary Dyskinesia
Brief Title: Glycine and Magnesium+Thiamine for the Treatment of Primary Ciliary Dyskinesia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Nacional de Enfermedades Respiratorias (Other Government)
Responsible Party: Principal Investigator, Mario H. Vargas, Senior Researcher, Instituto Nacional de Enfermedades Respiratorias
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C16-24
Record Dates: First submitted 2025-04-28; First posted 2025-05-06 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-10

CONDITIONS: Primary Ciliary Dyskinesia
Keywords: Primary ciliary dyskinesia; Glycine; Magnesium; Lung function; thiamine; benfotiamine
MeSH Terms: conditions — Ciliary Motility Disorders | interventions — Glycine

STUDY DESIGN:
Intervention Model Description: Four arms, parallel design, placebo controlled.
Who Masked: Participant, Care Provider
Masking Description: All study arms will receive similar bottles containing a whitish powder with the corresponding treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Glycine (Experimental): Patients will receive for 6 months an oral supplement of 0.5 g/kg/day glycine, up to 25 g/day, divided in three daily intakes.
  Interventions: Dietary Supplement: Glycine
- Magnesium+thiamine (Experimental): Patients will receive for 6 months an oral supplement of up to 400 mg/day, according to age, of elementary magnesium (formulated as magnesium citrate) plus up to 10 mg/day of thiamine (formulated as benfotiamine), divided in three daily intakes.
  Interventions: Dietary Supplement: Magnesium+thiamine
- Glycine plus magnesium+thiamine (Experimental): Patients will receive for 6 months oral supplements of glycine and magnesium+thiamine, as described.
  Interventions: Dietary Supplement: Glycine; Dietary Supplement: Magnesium+thiamine
- Placebo (Placebo Comparator): Patients will receive for 6 months placebo (sugar glass), in a similar daily amount as in experimental arms, and divided in three daily intakes.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Glycine — Patients will receive for 6 months an oral supplement of 0.5 g/kg/day glycine, up to 25 g/day, divided in three daily intakes.
  Arms: Glycine; Glycine plus magnesium+thiamine
Dietary Supplement: Magnesium+thiamine — Patients will receive for 6 months an oral supplement of up to 400 mg/day, according to age, of elementary magnesium (formulated as magnesium citrate) plus up to 10 mg/day of thiamine (formulated as benfotiamine), divided in three daily intakes.
  Arms: Glycine plus magnesium+thiamine; Magnesium+thiamine
Other: Placebo — Patients will receive for 6 months placebo (sugar glass), in a similar daily amount as in experimental arms, and divided in three daily intakes.
  Arms: Placebo

SUMMARY:
* Patients with primary ciliary dyskinesia (PCD) have trouble with clearing their bronchi from mucus, which in the long-term may produce severe damage to the lungs. Currently, there is no specific treatment for PCD beyond supportive measures such as airway hydration and postural drainage.
* Glycine is an amino acid with anti-inflammatory properties that proved to be beneficial in another disease with problematic airway clearance, cystic fibrosis.
* Magnesium participates in many crucial chemical reactions, including some that might favor fluidification and mobilization of mucus. Thiamine (vitamin B1) co-participates with magnesium in some mitochondrial enzymatic reactions occurring in the citric acid cycle.
* Thus, oral supplements of glycine and magnesium+thiamine might improve symptoms and lung function of patients with PCD, and these effects may even be better if these supplements are combined.
* In this study, in addition to their usual care, patients with PCD will receive for 6 months one of the following treatments: 1) an oral supplement of 0.5 g/kg/day glycine, 2) an oral supplement of up to 400 mg/day elementary magnesium plus up to 10 mg/day thiamine, according to the subject's age, 3) glycine plus magnesium+thiamine supplements, as described, or 4) a placebo, which is an inert substance. All treatments will be administered as a whitish powder contained in similar bottles.
* The investigators will evaluate whether glycine and/or magnesium+thiamine reduce exacerbations of the disease, improve pulmonary function and quality of life, and reduce some pro-inflammatory compounds measured in saliva.

DETAILED DESCRIPTION:
Background Primary ciliary dyskinesia (PCD) is characterized by ciliary dysfunction causing mucus accumulation in the airways that favors recurrent infections and bronchiectasis. Apart from general airway clearance, few therapeutic alternatives exist for PCD, and these are usually derived from experiences obtained from other lung diseases such as cystic fibrosis. Among the few clinical trials focused on PCD, the use of azithromycin for 6 months decreased the number of respiratory exacerbations, but with little or no impact on lung function or quality of life. Likewise, although useful in cystic fibrosis, inhalation of hypertonic saline and oral administration of N-acetylcysteine did not improve respiratory symptoms in patients with PCD. Therefore, it is urgent to find therapeutic approaches that prevent respiratory exacerbations, improve quality of life and, ideally, improve lung function. A lot of scientific literature supports the potential beneficial effect of glycine and/or magnesium+thiamine supplements in patients with PCD, as described below. Thus, in this study the investigators will evaluate the effect of glycine and magnesium+thiamine supplementation, alone or combined, in patients with PCD.

Characteristics of glycine Glycine is a non-essential and the simplest amino acid. Physically, it is a whitish powder with a sweet taste, soluble in water and relatively inexpensive (approximately $27 dollars per kg). Aside from participating in protein composition, glycine is an agonist for its own specific receptors (GlyR), which are chloride channels that cause membrane hyperpolarization. In excitable cells such as neurons, glycine is an inhibitory neurotransmitter, while in other cells such as Kupffer cells, alveolar macrophages and neutrophils, this amino acid reduces the sensitivity to proinflammatory stimuli. This stabilizing effect on inflammatory cells has been corroborated in several studies. For example, glycine decreases the expression and levels of tumor necrosis factor (TNF)-α and IL-6 in mouse adipose tissue and prevents the production of TNF-α and superoxide anion in lipopolysaccharide-stimulated alveolar macrophages, as well as TNF-α and IL-6 in 3T3-L1 cells, probably through the inhibition of IKK-α/β and, therefore, of NF-kB phosphorylation. In animal models of endotoxic shock, glycine protects from structural damage and decreases neutrophilic inflammation and proinflammatory cytokine production, probably through inhibition of NF-kB and NLRP3, as well as restoration of NRF2. Recently, in a controlled, crossover clinical trial the investigators administered 0.5 g/kg/day of glycine orally for 8 weeks to children with cystic fibrosis (Vargas et al. BMC Pulm Med 2017;17(1):206. doi: 10.1186/s12890-017-0528-x). This study demonstrated that glycine induced an improvement in clinical and spirometric variables, as well as a decrease in serum TNF-α and a trend towards a decrease in IL-6 and G-CSF. In this and many other studies, oral glycine was virtually devoid of adverse effects.

Possible role of magnesium and thiamine in PCD Epidemiological studies have shown that hypomagnesemia is highly prevalent in the general population, even among self-reported healthy individuals, being as high as 30%. This can be explained by several factors, including Western-type diet, decreased concentration of magnesium in vegetables, use of medications that decrease the intestinal absorption of magnesium or favor its renal elimination, and genetic variants of magnesium transport proteins. Therefore, in patients with PCD, it is expected that at least a similar percentage have a magnesium deficiency. In humans, magnesium is an indispensable element for the proper functioning of at least 300 enzymes involved in vital processes, including those involved in relevant intracellular signaling pathways, for example, kinases (which phosphorylate substrates from ATP-Mg2+), adenylate cyclase (which generates the second messenger cyclic AMP) and G proteins (key GTPases in intracellular signaling of many receptors). Therefore, a relative magnesium deficiency could affect the function of virtually any tissue. In addition, it has been shown that the activity of exogenous rhDNase or endogenous DNases require magnesium in the microenvironment. On the other hand, magnesium is an indispensable cofactor for ATP (ATP-Mg2+) to be utilized by the ATPase domain of dynein and to generate the ciliary beating movement. Therefore, magnesium is important also for mucous fluidification and ciliary functioning. Finally, one of the most relevant metabolic pathways where magnesium is essential is the citric acid cycle, which is the main energy (ATP) generator in the mitochondria, since it is a cofactor of pyruvate dehydrogenase, alpha-ketoglutarate dehydrogenase and branched-chain keto amino acid dehydrogenase, as well as other related enzymes such as transketolase and 2-hydroxyacyl CoA lyase. It is important to note that in addition to magnesium, all these enzymes also require thiamine diphosphate, so that the deficiency of either cofactor (magnesium and thiamine) leads to mitochondrial dysfunction. This is particularly relevant in PCD because proper mitochondrial function is essential for the formation and functioning of cilia.

Hypothesis

1. In patients with PCD, glycine or magnesium+thiamine supplementation for 6 months will be associated with a 25% decrease in the number of respiratory exacerbations compared to placebo.
2. In patients with PCD, combined glycine and magnesium+thiamine supplements for 6 months will be associated with a 50% decrease in the number of respiratory exacerbations compared to placebo.

Major objective To evaluate the effect of glycine and magnesium+thiamine supplements, alone or combined, administered for 6 months to patients with PCD on the number of respiratory exacerbations.

Secondary objectives

To evaluate the effect of glycine and magnesium+thiamine supplements, alone or combined, administered for 6 months to patients with PCD on:

1. Quality of life (questionnaire of the Spanish version of the QOL-PCD, as well as some questions on possible side effects).
2. Growth and development (weight-for-height, height-for-age, BMI).
3. Peripheral oxygen saturation (SpO2).
4. Pulmonary function tests (nasal nitric oxide, oscillometry, multiple breath nitrogen washout, spirometry, 6-min walking test).
5. Biomarkers in saliva (IL-1β, IL-6, IL-8, TNF-α, MPO).

Description of the study The study will be carried out at the Instituto Nacional de Enfermedades Respiratorias (INER), located in Mexico City. Once an informed consent is signed by patients or their legal guardians, participants will be randomly allocated to one of four study arms: 1) glycine, 2) magnesium+thiamine, 3) glycine and magnesium+thiamine, 4) placebo. Glycine will be administered at a dose of 0.5 g/kg/day, up to a maximum of 25 g/day. The dose of magnesium will be 8 mg/kg/day of elementary magnesium administered as magnesium citrate, up to a maximum of 400 mg/day. The dose of thiamine will be 0.2 mg/kg/day administered as benfotiamine, up to a maximum of 10 mg/day. Patients or their legal guardians will be asked to fill out an online symptom questionnaire every week. At the initial visit and every 2 months the following maneuvers will be performed: inquiry about pulmonary exacerbations; weight and height measurements; physical examination; pulse oximetry; saliva sampling for measuring IL-1β, IL-6, IL-8, TNF-α, myeloperoxidase (MPO) and albumin; nasal nitric oxide measurement; basal oscillometry; multiple breath nitrogen washout test; basal spirometry; post-salbutamol oscillometry and spirometry, 6-min walk test. In each visit, except for the final visit, a 500 g plastic bottle with a mixture of glycine, magnesium+thiamine, and/or placebo (sugar glass) powders, according to their assigned group, will be given to the patient or to the person at charge. All bottles will be identical in appearance.

Sample size Due to feasibility reasons, the investigators consider that the number of participants in each of the four groups will be n=15 (total n=60 patients).

ELIGIBILITY:
Inclusion Criteria:

1. Any sex.
2. Age of 5 years or more.
3. Diagnosis of primary ciliary dyskinesia (PCD) established according to international recommendations (Shapiro et al. Am J Respir Crit Care Med 2018;197(12):e24-e39, and Shapiro et al. Ped Pulmonol 2016;51:115-132).
4. Without respiratory exacerbations of PCD in the previous 30 days.
5. Without acute respiratory infection in the previous 30 days.
6. Informed consent letter signed by the patient (if the patient's age is 18 years or more).
7. Informed consent letter signed by the legal guardian, and assent letter signed by the patient (if the patient's age is <18 years).

Exclusion Criteria:

1. Participation in other research protocol involving therapeutic measures.

Elimination Criteria:

1. None.

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-10-02 (Actual); Primary Completion 2028-03 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Number of respiratory exacerbations | 6 months
  A respiratory exacerbation will be defined as: 1) any increase in respiratory symptoms that motivated the initiation of antibiotic therapy, or 2) a 10% or more decrease in FEV1 with respect to the FEV1 value at recruitment. A blinded pediatric pulmonologist will review all cases to corroborate whether a suspected episode was indeed a respiratory exacerbation.

SECONDARY OUTCOMES:
Quality of life-Primary ciliary dyskinesia questionnaire (QOL-PCD) | 6 months
  The quality of life will be assessed weekly by the Spanish version of the QOL-PCD questionnaire, as well as by some questions on possible side effects, filled online.
Weight-for-height | 6 months
  The z score of weight-for-height will be used as a proxy for assessing the child's growth and development every two months.
Height-for-age | 6 months
  The z score of height-for-age will be used as a proxy for assessing the child's growth and development every two months.
SpO2 | 6 months
  Peripheral blood oxygen saturation, as measured by pulse oximetry every two months.
Body mass index | 6 months
  The z score of body mass index will be used as a proxy for assessing the child's growth and development every two months
Nasal nitric oxide | 6 months
  The level (nL/min) of nasal nitric oxide measured every two months.
R5 | 6 months
  Respiratory system resistance in kPa/(L/s) measured every two months by impulse oscillometry at 5 Hz (a proxy of total airway resistance).
R20 | 6 months
  Respiratory system resistance in kPa/(L/s) measured every two months by impulse oscillometry at 20 Hz (a proxy of large airway resistance).
R5-R20 | 6 months
  Difference between respiratory system resistances at 5 and 20 Hz, measured every two months by impulse oscillometry (a proxy of peripheral airway resistance).
(R5-R20)/R5 | 6 months
  Difference between respiratory system resistances at 5 and 20 Hz, divided by R5, measured every two months by impulse oscillometry (a proxy of peripheral airway resistance).
X5 | 6 months
  Respiratory system reactance in kPa/(L/s) measured every two months by impulse oscillometry at 5 Hz (a proxy of lung parenchyma/peripheral airway status).
X20 | 6 months
  Respiratory system reactance in kPa/(L/s) measured every two months by impulse oscillometry at 20 Hz (a proxy of lung parenchyma/peripheral airway status).
Frequency of resonance (Fres) | 6 months
  Hz at which lung elastance and inertance are in equilibrium, as measured every two months by impulse oscillometry.
Area of reactance (AX) | 6 months
  Area, in kPa/L, limited below by X5 and Fres, and above by the zero reactance, as measured every two months by impulse oscillometry.
Multiple breath nitrogen washout | 6 months
  Lung clearance index measured every two months by multiple breath nitrogen washout.
FVC | 6 months
  Forced vital capacity, measured every two months by spirometry.
FEV1 | 6 months
  Forced expiratory volume at the first second, measured every two months by spirometry.
FEV1/FVC | 6 months
  Ratio of forced expiratory volume at the first second and forced vital capacity, measured every two months by spirometry.
Response to bronchodilator (oscillometry) | 6 months
  Change in lung function, as assessed by oscillometry, after the inhalation of a bronchodilator (salbutamol), measured every two months.
Response to bronchodilator (spirometry) | 6 months
  Change in lung function, as assessed by spirometry, after the inhalation of a bronchodilator (salbutamol), measured every two months.
6-minute walk test | 6 months
  Exercise test performed every two months in which the subject walks in a flat surface for 6 minutes to evaluate the maximum distance achieved.
IL-1beta in saliva | 6 months
  Interleukin 1 beta, measured in a saliva sample.
IL-6 in saliva | 6 months
  Interleukin 6, measured in a saliva sample.
IL-8 in saliva | 6 months
  Interleukin 8, measured in a saliva sample.
TNF-alpha in saliva | 6 months
  Tumor necrosis factor alpha, measured in a saliva sample.
MPO in saliva | 6 months
  Neutrophilic myeloperoxidase, measured in a saliva sample.

CONTACTS AND LOCATIONS:
Overall Officials: Mario H. Vargas, MSc, Principal Investigator — 5556665868
Locations (1):
- Instituto Nacional de Enfermedades Respiratorias, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: Yes
Data will be available upon reasonable request for research purposes.
Supporting Information: Study Protocol, CSR
Time Frame: Data will be available indefinitely after publication of the results.
Access Criteria: Reasonable request directed to the principal investigator.

REFERENCES:
- [Background] Piatti G, De Santi MM, Farolfi A, Zuccotti GV, D'Auria E, Patria MF, Torretta S, Consonni D, Ambrosetti U. Exacerbations and Pseudomonas aeruginosa colonization are associated with altered lung structure and function in primary ciliary dyskinesia. BMC Pediatr. 2020 Apr 13;20(1):158. doi: 10.1186/s12887-020-02062-4. PMID 32284045
- [Background] Sagel SD, Kupfer O, Wagner BD, Davis SD, Dell SD, Ferkol TW, Hoppe JE, Rosenfeld M, Sullivan KM, Tiddens HAWM, Knowles MR, Leigh MW. Airway Inflammation in Children with Primary Ciliary Dyskinesia. Ann Am Thorac Soc. 2023 Jan;20(1):67-74. doi: 10.1513/AnnalsATS.202204-314OC. PMID 35984413
- [Background] Gontijo-Amaral C, Guimaraes EV, Camargos P. Oral magnesium supplementation in children with cystic fibrosis improves clinical and functional variables: a double-blind, randomized, placebo-controlled crossover trial. Am J Clin Nutr. 2012 Jul;96(1):50-6. doi: 10.3945/ajcn.112.034207. Epub 2012 May 30. PMID 22648717
- [Background] Vargas MH, Del-Razo-Rodriguez R, Lopez-Garcia A, Lezana-Fernandez JL, Chavez J, Furuya MEY, Marin-Santana JC. Effect of oral glycine on the clinical, spirometric and inflammatory status in subjects with cystic fibrosis: a pilot randomized trial. BMC Pulm Med. 2017 Dec 15;17(1):206. doi: 10.1186/s12890-017-0528-x. PMID 29246256
- [Background] Kobbernagel HE, Buchvald FF, Haarman EG, Casaulta C, Collins SA, Hogg C, Kuehni CE, Lucas JS, Moser CE, Quittner AL, Raidt J, Rosthoj S, Sorensen AL, Thomsen K, Werner C, Omran H, Nielsen KG. Efficacy and safety of azithromycin maintenance therapy in primary ciliary dyskinesia (BESTCILIA): a multicentre, double-blind, randomised, placebo-controlled phase 3 trial. Lancet Respir Med. 2020 May;8(5):493-505. doi: 10.1016/S2213-2600(20)30058-8. PMID 32380069
- [Background] Paff T, Daniels JM, Weersink EJ, Lutter R, Vonk Noordegraaf A, Haarman EG. A randomised controlled trial on the effect of inhaled hypertonic saline on quality of life in primary ciliary dyskinesia. Eur Respir J. 2017 Feb 23;49(2):1601770. doi: 10.1183/13993003.01770-2016. Print 2017 Feb. PMID 28232410
- [Background] Jensen T, Kharazmi A, Schiotz PO, Nielsen H, Stenvang Pedersen S, Stafanger G, Koch C, Hoiby N. Effect of oral N-acetylcysteine administration on human blood neutrophil and monocyte function. APMIS. 1988 Jan;96(1):62-7. doi: 10.1111/j.1699-0463.1988.tb05269.x. PMID 3345250
- [Background] Jentsch TJ, Stein V, Weinreich F, Zdebik AA. Molecular structure and physiological function of chloride channels. Physiol Rev. 2002 Apr;82(2):503-68. doi: 10.1152/physrev.00029.2001. PMID 11917096
- [Background] Van den Eynden J, Ali SS, Horwood N, Carmans S, Brone B, Hellings N, Steels P, Harvey RJ, Rigo JM. Glycine and glycine receptor signalling in non-neuronal cells. Front Mol Neurosci. 2009 Aug 20;2:9. doi: 10.3389/neuro.02.009.2009. eCollection 2009. PMID 19738917
- [Background] Wheeler MD, Rose ML, Yamashima S, Enomoto N, Seabra V, Madren J, Thurman RG. Dietary glycine blunts lung inflammatory cell influx following acute endotoxin. Am J Physiol Lung Cell Mol Physiol. 2000 Aug;279(2):L390-8. doi: 10.1152/ajplung.2000.279.2.L390. PMID 10926563
- [Background] Alarcon-Aguilar FJ, Almanza-Perez J, Blancas G, Angeles S, Garcia-Macedo R, Roman R, Cruz M. Glycine regulates the production of pro-inflammatory cytokines in lean and monosodium glutamate-obese mice. Eur J Pharmacol. 2008 Dec 3;599(1-3):152-8. doi: 10.1016/j.ejphar.2008.09.047. Epub 2008 Oct 9. PMID 18930730
- [Background] Almanza-Perez JC, Alarcon-Aguilar FJ, Blancas-Flores G, Campos-Sepulveda AE, Roman-Ramos R, Garcia-Macedo R, Cruz M. Glycine regulates inflammatory markers modifying the energetic balance through PPAR and UCP-2. Biomed Pharmacother. 2010 Oct;64(8):534-40. doi: 10.1016/j.biopha.2009.04.047. Epub 2009 Oct 17. PMID 19864106
- [Background] Wheeler MD, Thurman RG. Production of superoxide and TNF-alpha from alveolar macrophages is blunted by glycine. Am J Physiol. 1999 Nov;277(5):L952-9. doi: 10.1152/ajplung.1999.277.5.L952. PMID 10564180
- [Background] Garcia-Macedo R, Sanchez-Munoz F, Almanza-Perez JC, Duran-Reyes G, Alarcon-Aguilar F, Cruz M. Glycine increases mRNA adiponectin and diminishes pro-inflammatory adipokines expression in 3T3-L1 cells. Eur J Pharmacol. 2008 Jun 10;587(1-3):317-21. doi: 10.1016/j.ejphar.2008.03.051. Epub 2008 Apr 8. PMID 18499099
- [Background] Contreras-Nunez E, Blancas-Flores G, Cruz M, Almanza-Perez JC, Gomez-Zamudio JH, Ventura-Gallegosc JL, Zentella-Dehesa A, Roberto-Lazzarini, Roman-Ramos R, Alarcon-Aguilar FJ. Participation of the IKK-alpha/beta complex in the inhibition of the TNF-alpha/NF-kappaB pathway by glycine: Possible involvement of a membrane receptor specific to adipocytes. Biomed Pharmacother. 2018 Jun;102:120-131. doi: 10.1016/j.biopha.2018.03.048. Epub 2018 Mar 22. PMID 29550635
- [Background] Ikejima K, Iimuro Y, Forman DT, Thurman RG. A diet containing glycine improves survival in endotoxin shock in the rat. Am J Physiol. 1996 Jul;271(1 Pt 1):G97-103. doi: 10.1152/ajpgi.1996.271.1.G97. PMID 8760112
- [Background] Zhang Y, Jia H, Jin Y, Liu N, Chen J, Yang Y, Dai Z, Wang C, Wu G, Wu Z. Glycine Attenuates LPS-Induced Apoptosis and Inflammatory Cell Infiltration in Mouse Liver. J Nutr. 2020 May 1;150(5):1116-1125. doi: 10.1093/jn/nxaa036. PMID 32101618
- [Background] Schimatschek HF, Rempis R. Prevalence of hypomagnesemia in an unselected German population of 16,000 individuals. Magnes Res. 2001 Dec;14(4):283-90. PMID 11794636
- [Background] Rodriguez-Ramirez M, Simental-Mendia LE, Gonzalez-Ortiz M, Martinez-Abundis E, Madero A, Brito-Zurita O, Perez-Fuentes R, Revilla-Monsalve C, Islas-Andrade S, Rodriguez-Moran M, Guerrero-Romero F. Prevalence of Prehypertension in Mexico and Its Association With Hypomagnesemia. Am J Hypertens. 2015 Aug;28(8):1024-30. doi: 10.1093/ajh/hpu293. Epub 2015 Jan 23. PMID 25618517
- [Background] Workinger JL, Doyle RP, Bortz J. Challenges in the Diagnosis of Magnesium Status. Nutrients. 2018 Sep 1;10(9):1202. doi: 10.3390/nu10091202. PMID 30200431
- [Background] Wolf FI, Cittadini A. Chemistry and biochemistry of magnesium. Mol Aspects Med. 2003 Feb-Jun;24(1-3):3-9. doi: 10.1016/s0098-2997(02)00087-0. No abstract available. PMID 12537985
- [Background] Birnbaumer L, Zurita AR. On the roles of Mg in the activation of G proteins. J Recept Signal Transduct Res. 2010 Dec;30(6):372-5. doi: 10.3109/10799893.2010.508165. Epub 2010 Aug 23. PMID 20731539
- [Background] Sanders NN, Franckx H, De Boeck K, Haustraete J, De Smedt SC, Demeester J. Role of magnesium in the failure of rhDNase therapy in patients with cystic fibrosis. Thorax. 2006 Nov;61(11):962-8. doi: 10.1136/thx.2006.060814. PMID 17071834
- [Background] Rosenecker J, Naundorf S, Rudolph C. Airway surface liquid contains endogenous DNase activity which can be activated by exogenous magnesium. Eur J Med Res. 2009 Jul 22;14(7):304-8. doi: 10.1186/2047-783x-14-7-304. PMID 19661013
- [Background] Warner FD, Mitchell DR. Dynein: the mechanochemical coupling adenosine triphosphatase of microtubule-based sliding filament mechanisms. Int Rev Cytol. 1980;66:1-43. doi: 10.1016/s0074-7696(08)61970-1. No abstract available. PMID 6446527
- [Background] Farrell PM, Fox GN, Spicer SS. Determination and characterization of ciliary ATPase in the presence of serum from cystic fibrosis patients. Pediatr Res. 1976 Feb;10(2):127-35. doi: 10.1203/00006450-197602000-00012. PMID 128730
- [Background] Ott M, Werneke U. Wernicke's encephalopathy - from basic science to clinical practice. Part 1: Understanding the role of thiamine. Ther Adv Psychopharmacol. 2020 Dec 29;10:2045125320978106. doi: 10.1177/2045125320978106. eCollection 2020. PMID 33447357
- [Background] Mrowicka M, Mrowicki J, Dragan G, Majsterek I. The importance of thiamine (vitamin B1) in humans. Biosci Rep. 2023 Oct 31;43(10):BSR20230374. doi: 10.1042/BSR20230374. PMID 37389565
- [Background] Pilchova I, Klacanova K, Tatarkova Z, Kaplan P, Racay P. The Involvement of Mg2+ in Regulation of Cellular and Mitochondrial Functions. Oxid Med Cell Longev. 2017;2017:6797460. doi: 10.1155/2017/6797460. Epub 2017 Jul 5. PMID 28757913
- [Background] Burkhalter MD, Sridhar A, Sampaio P, Jacinto R, Burczyk MS, Donow C, Angenendt M; Competence Network for Congenital Heart Defects Investigators; Hempel M, Walther P, Pennekamp P, Omran H, Lopes SS, Ware SM, Philipp M. Imbalanced mitochondrial function provokes heterotaxy via aberrant ciliogenesis. J Clin Invest. 2019 May 16;129(7):2841-2855. doi: 10.1172/JCI98890. PMID 31094706
- [Background] Satir P. Structural basis of ciliary movement. Environ Health Perspect. 1980 Apr;35:77-82. doi: 10.1289/ehp.803577. PMID 6447592
- [Background] Marthin JK, Petersen N, Skovgaard LT, Nielsen KG. Lung function in patients with primary ciliary dyskinesia: a cross-sectional and 3-decade longitudinal study. Am J Respir Crit Care Med. 2010 Jun 1;181(11):1262-8. doi: 10.1164/rccm.200811-1731OC. Epub 2010 Feb 18. PMID 20167855
- [Background] Lucas JS, Behan L, Dunn Galvin A, Alpern A, Morris AM, Carroll MP, Knowles MR, Leigh MW, Quittner AL. A quality-of-life measure for adults with primary ciliary dyskinesia: QOL-PCD. Eur Respir J. 2015 Aug;46(2):375-83. doi: 10.1183/09031936.00216214. Epub 2015 May 14. PMID 25976687
- [Background] Shapiro AJ, Davis SD, Polineni D, Manion M, Rosenfeld M, Dell SD, Chilvers MA, Ferkol TW, Zariwala MA, Sagel SD, Josephson M, Morgan L, Yilmaz O, Olivier KN, Milla C, Pittman JE, Daniels MLA, Jones MH, Janahi IA, Ware SM, Daniel SJ, Cooper ML, Nogee LM, Anton B, Eastvold T, Ehrne L, Guadagno E, Knowles MR, Leigh MW, Lavergne V; American Thoracic Society Assembly on Pediatrics. Diagnosis of Primary Ciliary Dyskinesia. An Official American Thoracic Society Clinical Practice Guideline. Am J Respir Crit Care Med. 2018 Jun 15;197(12):e24-e39. doi: 10.1164/rccm.201805-0819ST. PMID 29905515
- [Background] Shapiro AJ, Zariwala MA, Ferkol T, Davis SD, Sagel SD, Dell SD, Rosenfeld M, Olivier KN, Milla C, Daniel SJ, Kimple AJ, Manion M, Knowles MR, Leigh MW; Genetic Disorders of Mucociliary Clearance Consortium. Diagnosis, monitoring, and treatment of primary ciliary dyskinesia: PCD foundation consensus recommendations based on state of the art review. Pediatr Pulmonol. 2016 Feb;51(2):115-32. doi: 10.1002/ppul.23304. Epub 2015 Sep 29. PMID 26418604
- [Background] Sheng L, Cao W, Lin P, Chen W, Xu H, Zhong C, Yuan F, Chen H, Li H, Liu C, Yang M, Li X. Safety, Tolerability and Pharmacokinetics of Single and Multiple Ascending Doses of Benfotiamine in Healthy Subjects. Drug Des Devel Ther. 2021 Mar 9;15:1101-1110. doi: 10.2147/DDDT.S296197. eCollection 2021. PMID 33727798
- [Background] Amado F, Calheiros-Lobo MJ, Ferreira R, Vitorino R. Sample Treatment for Saliva Proteomics. Adv Exp Med Biol. 2019;1073:23-56. doi: 10.1007/978-3-030-12298-0_2. PMID 31236838
- [Background] Beydon N, Kouis P, Marthin JK, Latzin P, Colas M, Davis SD, Haarman E, Harris AL, Hogg C, Kilbride E, Kuehni CE, Marangu D, Nielsen KG, Pendergrast C, Robinson P, Rumman N, Rutter M, Walker WT, Ferkol T, Lucas JS. Nasal nitric oxide measurement in children for the diagnosis of primary ciliary dyskinesia: European Respiratory Society technical standard. Eur Respir J. 2023 Apr 20;61(4):2202031. doi: 10.1183/13993003.02031-2022. Print 2023 Apr. PMID 36822632
- [Background] Shapiro AJ, Dell SD, Gaston B, O'Connor M, Marozkina N, Manion M, Hazucha MJ, Leigh MW. Nasal Nitric Oxide Measurement in Primary Ciliary Dyskinesia. A Technical Paper on Standardized Testing Protocols. Ann Am Thorac Soc. 2020 Feb;17(2):e1-e12. doi: 10.1513/AnnalsATS.201904-347OT. PMID 31770003
- [Background] King GG, Bates J, Berger KI, Calverley P, de Melo PL, Dellaca RL, Farre R, Hall GL, Ioan I, Irvin CG, Kaczka DW, Kaminsky DA, Kurosawa H, Lombardi E, Maksym GN, Marchal F, Oppenheimer BW, Simpson SJ, Thamrin C, van den Berge M, Oostveen E. Technical standards for respiratory oscillometry. Eur Respir J. 2020 Feb 27;55(2):1900753. doi: 10.1183/13993003.00753-2019. Print 2020 Feb. PMID 31772002
- [Background] Robinson PD, Latzin P, Verbanck S, Hall GL, Horsley A, Gappa M, Thamrin C, Arets HG, Aurora P, Fuchs SI, King GG, Lum S, Macleod K, Paiva M, Pillow JJ, Ranganathan S, Ratjen F, Singer F, Sonnappa S, Stocks J, Subbarao P, Thompson BR, Gustafsson PM. Consensus statement for inert gas washout measurement using multiple- and single- breath tests. Eur Respir J. 2013 Mar;41(3):507-22. doi: 10.1183/09031936.00069712. Epub 2013 Feb 8. PMID 23397305
- [Background] Graham BL, Steenbruggen I, Miller MR, Barjaktarevic IZ, Cooper BG, Hall GL, Hallstrand TS, Kaminsky DA, McCarthy K, McCormack MC, Oropez CE, Rosenfeld M, Stanojevic S, Swanney MP, Thompson BR. Standardization of Spirometry 2019 Update. An Official American Thoracic Society and European Respiratory Society Technical Statement. Am J Respir Crit Care Med. 2019 Oct 15;200(8):e70-e88. doi: 10.1164/rccm.201908-1590ST. PMID 31613151
- [Background] Holland AE, Spruit MA, Troosters T, Puhan MA, Pepin V, Saey D, McCormack MC, Carlin BW, Sciurba FC, Pitta F, Wanger J, MacIntyre N, Kaminsky DA, Culver BH, Revill SM, Hernandes NA, Andrianopoulos V, Camillo CA, Mitchell KE, Lee AL, Hill CJ, Singh SJ. An official European Respiratory Society/American Thoracic Society technical standard: field walking tests in chronic respiratory disease. Eur Respir J. 2014 Dec;44(6):1428-46. doi: 10.1183/09031936.00150314. Epub 2014 Oct 30. PMID 25359355